CLINICAL TRIAL: NCT07350369
Title: Research on Early Warning and Diagnosis & Treatment Pathway for Micro Kidney Stones
Status: Recruiting | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY20252397-F-1
Record Dates: First submitted 2025-12-25; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-10

CONDITIONS: Kidney Stone
MeSH Terms: conditions — Kidney Calculi | interventions — Blood Specimen Collection; Urination

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Nephrolithiasis: For eligible subjects who meet the inclusion and exclusion criteria, one tube (approximately 4 mL each) of blood and urine samples collected prior to surgery during hospitalization and already tested will be gathered. Serum will be separated from the blood samples, while the entire urine sample will be submitted without processing. These samples will undergo further targeted metabolomics analysis. By measuring amine-related substances using targeted metabolomics, differences in amine compounds and metabolites in blood and urine between kidney stone patients and healthy individuals will be analyzed.
  Interventions: Other: Detect the levels of metabolites in blood and urine
- Normal: For eligible subjects who meet the inclusion and exclusion criteria, one tube (approximately 4 mL each) of blood and urine samples collected prior to surgery during hospitalization and already tested will be gathered. Serum will be separated from the blood samples, while the entire urine sample will be submitted without processing. These samples will undergo further targeted metabolomics analysis. By measuring amine-related substances using targeted metabolomics, differences in amine compounds and metabolites in blood and urine between kidney stone patients and healthy individuals will be analyzed.
  Interventions: Other: Detect the levels of metabolites in blood and urine

INTERVENTIONS:
Other: Detect the levels of metabolites in blood and urine — Detect the levels of metabolites in blood and urine

SUMMARY:
Exploring abnormal metabolism in kidney stone patients and developing drugs for kidney stone treatment and their mechanisms of action.

DETAILED DESCRIPTION:
For eligible subjects who meet the inclusion and exclusion criteria, one tube (approximately 4 mL each) of blood and urine samples collected prior to surgery during hospitalization and already tested in clinical laboratories will be gathered. Serum will be separated from the blood samples, while the entire urine sample will be submitted without processing, for further targeted metabolomics analysis. By analyzing the results of targeted metabolomic profiling of amine-related substances, differences in amines and metabolites in blood and urine between kidney stone patients and healthy individuals will be assessed.

By measuring and comparing the levels of amine compounds in blood and their corresponding metabolites in urine, statistical analysis will be performed to identify specific amines that are elevated in blood and whose metabolites are simultaneously increased in urine. The underlying mechanisms of these elevations will be further investigated through experimental studies.

ELIGIBILITY:
Inclusion Criteria Case Group

* Inpatients treated in the Department of Urology at Xijing Hospital with a diagnosis of renal calculi confirmed by imaging examinations, including abdominal plain radiography, ultrasonography, or computed tomography (CT).
* Aged between 18 and 70 years, regardless of sex.
* Willing to participate in the study and providing informed consent for the use of residual blood and urine samples (remaining after routine clinical testing) for research purposes.
* Complete medical records available, including medical history, clinical symptoms, physical examination findings, previous treatments, and other relevant information.

Control Group

* Inpatients treated in the Department of Urology at Xijing Hospital with no evidence of kidney stones or other urological diseases, as confirmed by urinary system ultrasonography, abdominal plain radiography, or urinary CT.
* Aged between 18 and 70 years, with sex distribution matched to the case group.
* Willing to participate in the study and providing informed consent for the use of residual blood and urine samples (remaining after routine clinical testing) for research purposes.
* No history of kidney stones or other urological diseases.

Exclusion Criteria

* Presence of severe systemic diseases that may affect kidney stone formation, including malignant tumors, heart failure, liver failure, or renal failure (serum creatinine > 354 μmol/L).
* Presence of other urological diseases, such as pyelonephritis, renal tuberculosis, renal cysts, or renal tumors.
* Presence of endocrine disorders, including hyperparathyroidism or hyperadrenocorticism.
* Pregnant or lactating women.
* Patients with psychiatric disorders, individuals unable to cooperate with the study, or those with a history of substance abuse or alcoholism.
* History of surgical intervention or extracorporeal shock wave lithotripsy (ESWL) for kidney stones within the past 3 months.
* Current use of medications that may influence kidney stone formation (e.g., diuretics, vitamin D, or calcium supplements) and inability to discontinue these medications.
* Insufficient blood or urine sample volume to meet analytical requirements, or samples that were severely contaminated or of poor quality and unsuitable for analysis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged between 18 and 70 years, with or without kidney stones.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-01-01 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Using liquid chromatography to measure the levels of 21 neurotransmitters and 5 biogenic amines in the blood, as well as 51 gut microbiota-derived metabolites in the urine, of patients with kidney stones and those without. | 25.08.01-25.11.01
  Blood and urine samples were collected from kidney stone patients and non-stone controls. Absolute concentrations of 21 neurotransmitters (e.g., dopamine, L-tyrosine, serotonin, 5-HIAA, tyramine) and 5 biogenic amines (spermidine, spermine, putrescine, ornithine, arginine) in blood, and 51 gut microbiota-derived metabolites (e.g., uric acid, shikimic acid, L-tryptophan, indoxyl-β-D-glucoside, 4-hydroxyphenylacetic acid, etc.) in urine were quantified using liquid chromatography.
  All concentrations are reported in ng/g. Statistical analyses compared metabolite levels between groups and assessed their associations with kidney stone disease.

CONTACTS AND LOCATIONS:
Overall Officials: zhang ke ying zhang, doctor, Principal Investigator — 中国人民解放军空军军医大学第一附属医院
Locations (1):
- The First Affiliated Hospital of Air Force Medical University of the Chinese People's Liberation Army, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No